CLINICAL TRIAL: NCT01769807
Title: Effects of CPAP on Nitrate and Norepinephrine Levels in Severe and Mild-moderate Sleep Apnea
Brief Title: Efficacy Study of CPAP on Nitrate and Norepinephrine Levels in Severe and Mild-moderate Sleep Apnea (SABIO)
Acronym: SABIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Paula Pinto, PhD, University of Lisbon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEDOC; Fundação Ciência e Tecnologia (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia (FCT))
Record Dates: First submitted 2012-11-17; First posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep apnea; CPAP treatment; Plasma nitrate; Urinary norepinephrine; Blood pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPAP treatment (Experimental): 67 consecutive male patients with OSA were recruited: 36 with mild-moderate OSA and 31 with severe OSA. Data were collected in all subjects at baseline and after 1 month of CPAP.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — CPAP adaptation was performed by a sleep technician and the patients were instructed to use this for 1 month.
  Other Names: Automated pressure setting device (AutoSet Spirit, ResMed)

SUMMARY:
Reduced plasma nitrate (NOx) levels and increased urinary norepinephrine (U-NE) levels have been described in severe obstructive sleep apnea (OSA), and are reverted by continuous positive airway pressure (CPAP). The investigators wanted to know the effect of CPAP on these biomarkers in mild-moderate OSA.

DETAILED DESCRIPTION:
The investigators aimed to compare NOx and U-NE levels and blood pressure (BP) between male patients with mild-moderate and severe OSA and determine the impact of 1 month of CPAP therapy on these parameters.

The investigators undertook a prospective study of 67 consecutive OSA patients (36 mild-moderate, 31 severe). Measurements of plasma NOx at 11 pm, 4 am and 7 am, 24-h U-NE and ambulatory BP were obtained at baseline and after 1 month of CPAP.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of obstructive sleep apnea

Exclusion Criteria:

* current smoker
* respiratory disease
* cardiac disease (except for arterial hypertension)
* renal disorder
* hepatic disorder
* psychiatric disorder
* diabetes mellitus
* dyslipidemia
* rhinitis
* sinusitis
* acute illness
* daytime hypoxemia or hypercapnia
* therapy with oral nitrates
* therapy with angiotensin-converting enzyme inhibitors
* therapy with beta-blockers
* therapy with statins
* therapy with non-steroidal anti-inflammatory drugs
* presence of central respiratory events
* previous CPAP therapy
* previous uvulopalatopharyngoplasty

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2004-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Plasma nitrate (NOx) levels | one month
  After sleep apnea diagnosis, measurements of plasma NOx at 11 pm, 4 am and 7 am were obtained at baseline and after 1 month of CPAP.

SECONDARY OUTCOMES:
24 h Blood pressure | one month after CPAP
  Ambulatory BP were obtained at baseline and after 1 month of CPAP.
Urinary norepinephrine (U-NE) levels | One month
  After sleep apnea diagnosis, measurements of urinary norepinephrine levels were obtained at baseline and after 1 month of CPAP.

CONTACTS AND LOCATIONS:
Overall Officials: Paula G Pinto, PhD, Principal Investigator — University of Lisbon
Locations (1):
- Hospital Pulido Valente, Lisbon, Lisbon District, Portugal

REFERENCES:
- [Derived] Pinto P, Barbara C, Montserrat JM, Patarrao RS, Guarino MP, Carmo MM, Macedo MP, Martinho C, Dias R, Gomes MJ. Effects of CPAP on nitrate and norepinephrine levels in severe and mild-moderate sleep apnea. BMC Pulm Med. 2013 Mar 13;13:13. doi: 10.1186/1471-2466-13-13. PMID 23497046